CLINICAL TRIAL: NCT04830228
Title: BIOTRONIK Dynetic-35 for the Treatment of Peripheral Iliac Lesions, Using the Cobalt Chromium Balloon-expandable Dynetic-35 Stent in Association With Passeo-35 Xeo Peripheral Dilation Catheter
Brief Title: BIOTRONIK Dynetic-35 Stent for the Treatment of Peripheral Iliac Lesions
Acronym: BIONETIC-I
Status: Active, not recruiting | Type: Observational
Sponsor: Biotronik AG (Industry)
Responsible Party: Sponsor
Other Study IDs: C1903
Record Dates: First submitted 2021-03-31; First posted 2021-04-05 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Peripheral Artery Disease
Keywords: Iliac arteries
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Ballon expandable stent and PTA — Endovascular treatment for the peripheral artery disease of the Iliac artery

SUMMARY:
BIOTRONIK cobalt chromium balloon-expandable Dynetic-35 stent in association with Passeo-35 Xeo peripheral dilation catheter for the treatment of peripheral iliac lesions

DETAILED DESCRIPTION:
Prospective, international, multi-center, single-arm study with up to 60 months follow up to evaluate safety and effectiveness of BIOTRONIK's Dynetic-35 stent associated with the use of Passeo-35 Xeo for the treatment of peripheral artery disease (PAD) in subjects with atherosclerotic disease in iliac arteries

ELIGIBILITY:
Inclusion Criteria

1. Subject is ≥ 18 years or the minimum age required for legal adult consent in the country of enrolment
2. Subject is capable (no legally authorized representative allowed) to provide written informed consent as approved by the Institutional Review Board (IRB)/Ethics Committee (EC) of the respective clinical site prior to any study related procedure
3. Subject has provided written informed consent before any study specific test or procedure and is willing to comply with all protocol and follow-up requirements
4. De novo, restenotic or occluded lesion(s) representing atherosclerotic lesion(s) in the iliac arteries
5. Reference lumen (vessel) diameter between 5mm and 10mm
6. The target lesion can be successfully crossed with a guide wire
7. The target lesion length is ≤ 100 mm
8. Subjects has more than 70% stenosis in target lesion
9. Subject has an evidence of a patent profunda femoris or superficial femoral artery in the target limb
10. Subject has symptomatic iliac artery occlusive disease defined as Rutherford category 2 or higher eligible for stenting

Exclusion Criteria

1. Subject is pregnant and/or breastfeeding or planning to become pregnant during the course of the study.
2. Subject is with a current medical condition with a life expectancy of less than one year.
3. Pre-existing target iliac artery aneurysm or perforation or dissection
4. Any medical condition that in the opinion of the investigator poses an unacceptable risk for implant of a stent according to the study indications like, sensitivity to metal ions, intolerance to contrast or antiplatelet, anticoagulant or thrombolytic medications required per the protocol
5. Abdominal aortic aneurysm (AAA) contiguous to the iliac artery target lesion requiring treatment
6. The subject is currently participating in an investigational drug, biologic, or another device study and has not reached their primary endpoint yet
7. Refuses blood transfusion
8. Chronic renal insufficiency (Serum creatinine >2.5 mg/dL within 30 days prior to index procedure)
9. Subject has IFU listed contraindication(s)
10. Subject has in-stent restenosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll subjects who have peripheral artery disease (PAD) requiring endovascular treatment of de-novo, restenotic and in-stent atherosclerotic lesions in iliac arteries
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
MAE at 12 months post-index procedure. | 12 Months
  The MAE includes device or procedure related death within 30 days post index procedure, cdTLR, and major index limb amputation up to 12 months post index procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Brodmann, Prof. Dr., Principal Investigator — Substitute Head of the Clinical Division of Angiology, Department of Internal Medicine
Locations (15):
- LKH Univ.-Klinikum Graz, Ambulanz für Angiologie, Graz, Austria
- Belgium (4):
  - Zol Genk, Genk
  - UZ Gent, Ghent
  - Regionaal Ziekenhuis Heilig Hart Tienen, Tienen
  - Az Jan Potaels Vilvoorde, Vilvoorde
- France (2):
  - Hôpital Privé du grand Narbonne, Narbonne
  - Hôpital Ambroise Paré, Paris
- Germany (6):
  - Klinikum Bayreuth, Bayreuth
  - Universitätsklinikum Essen, Essen
  - Diakonissenkrankenhaus, Flensburg
  - Universitätsklinikum Jena, Jena
  - St. Franziskushospital Münster, Münster
  - Universitätsklinikum Tübingen, Tübingen
- Semmelweis University Hospital, Budapest, Hungary
- Pauls Stradins Clinical University Hospital, Riga, Latvia

REFERENCES:
- [Derived] Brodmann M, Nemes B, Moreels N, Austermann M, Schmehl J, Robijn J, Rammos C, Muller-Hulsbeck S, Keirse K, Coscas R, Kupcs K, Augustin AM, Moebius-Winkler S, Lichtenberg M, Lansink W. Dynetic-35 cobalt chromium balloon-expandable stent for iliac lesions: 12-month results of the BIONETIC-I multi-center study. CVIR Endovasc. 2025 Dec 13;8(1):114. doi: 10.1186/s42155-025-00633-z. PMID 41389246